CLINICAL TRIAL: NCT05973409
Title: Evaluation of Onefit Scleral Lenses in the Mangement of Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SEC-P052021
Record Dates: First submitted 2023-03-23; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: At the fitting visit, only uncoated lenses will be used to determine the parameters of the lenses to be ordered. At both dispense visits, participants and investigators will be masked to the lens type dispensed. In order to achieve this, unmasked study personnel will determine the order of lens wear according to the randomization schedule and they will not share the lens labels or packs with the investigator. Instead, the lenses will be transferred to an unmarked case/container prior to being provided at the Dispense visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Habitual Soft Lens Wearers (Experimental): Each group will be a prospective, randomized, double masked, cross-over, 1-month per arm, daily wear study. Each participant will be active in the study for at least 2 months.
  Interventions: Device: scleral lens
- Non Contact Lens Wearers (Experimental): Each group will be a prospective, randomized, double masked, cross-over, 1-month per arm, daily wear study. Each participant will be active in the study for at least 2 months.
  Interventions: Device: scleral lens

INTERVENTIONS:
Device: scleral lens — scleral lens with and without hydra-peg coating

SUMMARY:
This study is being conducted to determine if scleral lenses coated with Hydra-PED improve comfort and dryness.

DETAILED DESCRIPTION:
The objective of the study is to determine if scleral lenses with and scleral lenses without Hydra-PEG coating provide positive improvement in ocular comfort and dryness scores.

The effect of the study lenses and the coating, will be compared in a group of symptomatic soft lens wearers, and also in a group of symptomatic non contact lens wearers.

The primary outcome variable for this study is "overall ocular comfort" reported at the screening visit for the habitual vision correction, and at the 4-week follow-up visits for each of the two study lenses. using a 0-10 scale (0.5 steps).

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 17 years of age and have full legal capacity to volunteer;
2. Have read and signed an information consent letter;
3. Are willing and able to follow instructions and maintain the appointment schedule;
4. Agree to wear the study scleral lenses for at least 8 hours per day, 5 days a week;
5. Have a refraction between +20.00 and -20.00D and spectacle astigmatism of no more than -3.00DC in each eye;
6. Have best corrected visual acuity of 20/40 or better in each eye with the study lenses;
7. Demonstrate an acceptable fit with the study lenses;
8. Have no active ocular disease or inflammation;
9. Group 1: Habitual wearer of frequent replacement or daily disposable soft lenses;
10. Group 2: Have not worn contact lenses for 6 months;
11. Group 1: Contact lens wearers should score ≥12 on CLDEQ-8;
12. Group 2: Non contact lens wearers should score ≥13 on OSDI.

Exclusion Criteria:

1. Are participating in any concurrent clinical or research study, or have done so within the past 30 days;
2. Cannot achieve a successful lens fit or vision with the study lens;
3. Have been diagnosed with keratoconus or corneal distortion;
4. Have any known active* ocular condition, disease and/or infection;
5. Have a systemic or ocular condition that in the opinion of the investigator may affect a study outcome variable e.g. pingueculae;
6. Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
7. Group 2: Non-contact lens wearers who score ≥33 on OSDI and also demonstrate either corneal staining ≥3 (Oxford scale) or non-invasive tear break-up time ≤3 seconds#;
8. Have known sensitivity to the diagnostic sodium fluorescein to be used in the study;
9. Are pregnant, lactating or planning a pregnancy^ at the time of enrolment, by self report;
10. Have undergone refractive error surgery;
11. Are listed on the Delegation Log for this study.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
overall ocular comfort | 4 weeks
  reported at the screening visit for the habitual vision correction, and at the 4-week follow-up visits for each of the two study lenses. using a 0-10 scale (0.5 steps)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, Principal Investigator — Director, Centre for Ocular Research and Education
Locations (1):
- School of Optometry & Vision Sciences, Waterloo, Ontario, Canada